CLINICAL TRIAL: NCT02404857
Title: A Novel BCI-controlled Pneumatic Glove System for Neurorehabilitation Post-stroke
Brief Title: BCI Post-stroke Neurorehabilitation
Acronym: BCI-stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Université Montpellier (Other); National University of Ireland, Maynooth (Other); Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 9431
Record Dates: First submitted 2015-01-12; First posted 2015-04-01 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Poststroke/CVA Hemiparesis; Paralytic Stroke; Hand Flaccid Paralysis
Keywords: Post stroke; BCI; Reeducation; Hand movement
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chronic post-stroke (Experimental): Patients >6 months post-stroke with little to no hand movement. use of EEG based BCI in the neurorehabilitation process
  Interventions: Device: EEG based Brain Computer Interface

INTERVENTIONS:
Device: EEG based Brain Computer Interface — Using EEG signals to classify brain activity being 'rest' or 'active' to control the attached pneumatic glove and close the sensory-motor loop between intentional/mental movement and physical (though passive) movement.

SUMMARY:
The goal is to evaluate the potential of a EEG based BCI (Brain-Computer-Interface) connected to a non-invasive pneumatic glove for rehabilitation of hand-movements post-stroke.

DETAILED DESCRIPTION:
Brain computer interfaces (BCI) encompasses the usage of the brain signals to compensate for lost physical function. The current protocol evaluates the therapeutic potential of a EEG based driven BCI that is connected to a non-invasive pneumatic glove for rehabilitation of hand flexion/extension post-stroke. The system non-invasive, portable and low-cost. The utility and usability of the system will be investigated at two levels. First by means of questionnaires for patients and therapist and second by means of in depth analysis of the EEG signals during intended, imagined and passive driven hand movements in relation to no movement at all and the capacity of the BCI to distinguish between these conditions.

ELIGIBILITY:
Inclusion Criteria:

* > 6 months post-stroke (chronic), unilateral
* > 18 yrs
* little to no hand movement
* spasticity < 3 on modified Ashworth Scale

Exclusion Criteria:

* major cognitive deficits (Folstein mini mental status > 23
* strong hemi-neglect (Catherine Bergego scale > 15/30)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Performance of the BCI-system (evaluation of performance through patient questionaires & the performance of the BCI classifier during intended and imagined hand movements) | During the whole study. Assesment is made for each patient after his participation ( 2 hours).
  Evaluation of the BCI-platform performance through patient questionnaires & the performance of the BCI classifier during intended and imagined hand movements.

SECONDARY OUTCOMES:
EEG sensory-motor rhythm signals (Detailed analysis of the EEG signals in relation to the severity of the paresis and movement condition) | During the whole studyAssesment is made for each patient after his participation ( 2 hours).
  Detailed analysis of the EEG signals in relation to the severity of the paresis and movement condition

CONTACTS AND LOCATIONS:
Overall Officials: Liesjet Van Dokkum, PhD, Principal Investigator — CHRU Montpellier, Lapeyronie // Euromov-M2H, Montpellier University
Locations (1):
- CHRU Lapeyronie, Montpellier, Herault, France